CLINICAL TRIAL: NCT00417547
Title: Comparison of Body Dissatisfaction Among Islamic Veil Practicing (IVP), Non-Complete IVP, and Inconsiderate to IVP Women
Status: Completed | Type: Observational
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Dr Reza Rastmanesh, SBMU
Other Study IDs: NNFTRI
Record Dates: First submitted 2006-12-29; First posted 2007-01-01 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Depression; Body Dissatisfaction; Obesity; Eating Disorders
Keywords: Self Concept; Eating Disorder; Body Mass Index; Dressing; Islamic Veil
MeSH Terms: conditions — Depression; Obesity; Feeding and Eating Disorders

SUMMARY:
The aim of this research is to examine the social, psychological and Islamic veil practicing (IVP), non-complete IVP and Inconsiderate to IVP correlates of body mass index (BMI) status in a women population. It is hypothesized that women who are IVP would differ on depression, and social variables compared with their non-practicing peers.

DETAILED DESCRIPTION:
In this cross-sectional study, a population-based sample of 1774 female responded anonymously to an aerobic health club administered questionnaire. Body mass index was calculated from height and weight and categorized into four classes of underweight, normal, overweight, and obese. The questionnaire also included questions about social experiences, body dissatisfaction as Body Shape Questionnaire (BSQ), future goals and Islamic Veil Practicing (IVP). Persian version of Beck Depression Inventory (BDI-II Persian) and Rosenberg Self Esteem Scale was also distributed among six groups of women having IVP/regular exercise (RE), IVP/non-RE, Non-complete IVP/RE, Non-complete IVP/non-RE, Inconsiderate to IVP/RE, and Inconsiderate to IVP/non-RE. Correlations of BMI with social, psychological, future goals and IVP were explored

ELIGIBILITY:
Inclusion Criteria:

* Open for all women practicing Islamic veil, Non-complete IV, or Inconsiderate to IV

Exclusion Criteria:

* Overt signs of Anorexia Nervosa, Bulimia Nervosa

Ages: 12 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000
Dates: Start 2006-02; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: REZA RASTMANESH, Ph.D., Study Chair — Shahid Beheshti University of Medical Sciences
Locations (1):
- Aerobic Health Clubs, Tehran, Tehran Province, Iran

REFERENCES:
- [Result] Rastmanesh R, Gluck ME, Shadman Z. Comparison of body dissatisfaction and cosmetic rhinoplasty with levels of veil practicing in Islamic women. Int J Eat Disord. 2009 May;42(4):339-45. doi: 10.1002/eat.20613. PMID 19115373